CLINICAL TRIAL: NCT06083298
Title: Comparison Between Multifidus Cervicis and Inter-semispinal Plane Blocks in Analgesia After Cervical Spine Surgery: A Randomized Controlled Trial
Brief Title: Multifidus Cervicis and Inter-Semispinal Plane Blocks in Analgesia After Cervical Spine Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Shereen Elsayed Abd Ellatif, associate professor of anesthesia and surgical intensive care, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 10952//15-8-2023
Record Dates: First submitted 2023-10-08; First posted 2023-10-13 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Cervical Spine Surgery
Keywords: Multifidus Cervicis plane block; Inter-Semispinal Plane Block; analgesia
MeSH Terms: conditions — Agnosia | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Triple (Participant, Investigator, Outcomes Assessor)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- control group (Placebo Comparator): patients will be operated under general anesthesia
  Interventions: Procedure: control group
- MCP group (Active Comparator): patients will receive MCP block followed by general anesthesia
  Interventions: Procedure: MCP group
- ISP group (Active Comparator): patients will receive ISP block followed by general anesthesia
  Interventions: Procedure: ISP group

INTERVENTIONS:
Procedure: control group — patients will be operated under general anesthesia
  Arms: control group
Procedure: MCP group — patients will receive ultrasound-guided MCP block with 15 ml of bupivacaine 0.25% on each side followed by general anesthesia.
  Arms: MCP group
Procedure: ISP group — patients will receive ultrasound-guided ISP block with 15 ml of bupivacaine 0.25% on each side followed by general anesthesia.
  Arms: ISP group

SUMMARY:
Major spine surgery with multilevel instrumentation is followed by a large amount of opioid consumption, significant pain, and difficult mobilization Pain is one of the main factors limiting ambulation, increasing the risk of thromboembolism by immobility, and causing metabolic changes that affect other systems. Therefore, individualized pain management with the use of appropriate analgesic techniques is of paramount importance. Moreover, early intervention in rehabilitation aiming at a better postoperative recovery may reduce the length of hospital stay and return to daily activity. Effective pain management is one of the crucial components in enhanced recovery after surgery (ERAS).

Numerous regional anesthetic techniques have been used to provide analgesia following cervical spine surgery, including patient-controlled epidural analgesia, cervical paravertebral block, cervical plexus block, cervical erector spinae plane blocks, and local inﬁltration analgesia, however, each of these techniques has specific limitations that prevent them from being the analgesic technique of choice for such surgeries.

Up to the author's knowledge, there is no study done to compare multifidus cervicis plane block versus inter-semispinal plane block in a randomized controlled clinical trial as preemptive analgesia in patients undergoing cervical spine surgery.

DETAILED DESCRIPTION:
Spine surgeries are commonly associated with severe postoperative pain, particularly complex procedures such as laminectomy on more than two disc levels, or scoliosis surgery, especially on the first postoperative day. Spinal foraminal stenosis and disc herniation, occurring often around C5-C7 levels, are the most popular underlying pathologies of the cervical spine.

One of the keys to a patient's recovery following cervical spine surgery is effective postoperative pain management. Nowadays, the concept of pain management with multimodal analgesia and regional anesthesia plays a crucial role in postoperative analgesia reducing opioid consumption and improving early mobilization. Numerous regional anesthetic techniques have been used, including patient-controlled epidural analgesia, cervical paravertebral block, cervical plexus block, cervical erector spinae plane blocks, and local inﬁltration analgesia. However, some of these techniques have specific limitations that prevent them from being the analgesic technique of choice for cervical spine surgery, and the others are still under research for its effectiveness.

Several new paraspinal blocks have been described in the thoracic and lumbar regions in which the dorsal rami of cervical nerves can be blocked without the block needle entering the paravertebral space. Moreover, novel cervical region blocks, including cervical interfascial plane (CIP) block, multifidus cervicis plane block (MCP), inter-semispinal plane (ISP) block, and retrolaminar cervical block have been developed. All these interfascial plane blocks are considered as promising alternatives to neuraxial blockade for various surgeries.

Multifidus cervicis plane (MCP) block First described by Ohgoshi et al. as a case report for analgesia after cervical laminoplasty, where the local anesthetic was injected between the multifidus cervicis and semispinalis cervicis muscles fascial planes at C5 level. Furthermore, MCP block was effective in another study as a treatment for cervicogenic headaches.

The inter-semispinal plane (ISP) block is also described by Ohgoshi et al., by injecting local anesthetic into the fascial plane between the semispinalis cervicis and capitis muscles and it effectively blocked multiple dorsal rami of the cervical spinal nerves in healthy volunteers.

This study will be designed for evaluation and comparison between Multifidus cervicis and inter-semispinal plane blocks as pre-emptive analgesia for patients undergoing cervical spine surgery under general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Patient acceptance.

  * Age 21-60 years old.
  * BMI ≤ 30 kg/m2
  * ASA I - II.
  * Elective posterior cervical spine surgery under general anesthesia.

Exclusion Criteria:

* History of allergy to the LA agents used in this study

  * Skin lesion at the needle insertion site,
  * Those with bleeding disorders, sepsis, liver disease, and psychiatric disorders
  * History of chronic pain and taking analgesics
  * History of cognitive dysfunction or mental illness

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 105 (Estimated)
Dates: Start 2023-10-20 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
changes in Visual analogue scale (VAS)score | measured at 1 hour, 3 hours,6 hours,12hours,18hours, 24 hours postoperatively
  On a scale of 0-10, the patient will learn to quantify postoperative pain where 0= No pain and 10= Maximum worst pain

SECONDARY OUTCOMES:
Total dose of rescue analgesia | in the first 24 hour postoperatively
  once the VAS score will be ≥ 3, rescue analgesia in the form of 0.1 mg/kg nalbuphine will be given and the total dose consumed will be recorded
the first time to rescue analgesia | in the first 24 hour postoperatively
  the time from the end of operation to patient reporting VAS ≥ 3

CONTACTS AND LOCATIONS:
Overall Officials: Shereen E Abd Ellatif, MD, Principal Investigator — Faculty of medicine, zagazig university
Locations (1):
- Faculty of medicine, zagazig university, Zagazig, Alsharqia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
planned after the completion of the study and publication
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: planned after the completion of the study and publication
Access Criteria: contact with the principal investigator

REFERENCES:
- [Background] Ohgoshi Y, Izawa H, Kori S, Matsukawa M. Multifidus cervicis plane block is effective for cervical spine surgery. Can J Anaesth. 2017 Mar;64(3):329-330. doi: 10.1007/s12630-016-0767-y. Epub 2016 Nov 3. No abstract available. PMID 27812925
- [Background] Ohgoshi Y, Nishizakura R, Takahashi Y, Takeda K, Nakayama H, Kawamata M, Kurahashi K. Novel ultrasound-guided inter-semispinal plane block: a comparative pilot study in healthy volunteers. J Anesth. 2018 Feb;32(1):143-146. doi: 10.1007/s00540-017-2439-7. Epub 2017 Dec 21. PMID 29270836
- [Background] Mostafa SF, Abu Elyazed MM, Eid GM, Belal AM. Inter-semispinal plane (ISP) block for postoperative analgesia following cervical spine surgery: A prospective randomized controlled trial. J Clin Anesth. 2022 Dec;83:110974. doi: 10.1016/j.jclinane.2022.110974. Epub 2022 Oct 10. PMID 36228453
- [Background] Hand WR, Taylor JM, Harvey NR, Epperson TI, Gunselman RJ, Bolin ED, Whiteley J. Thoracolumbar interfascial plane (TLIP) block: a pilot study in volunteers. Can J Anaesth. 2015 Nov;62(11):1196-200. doi: 10.1007/s12630-015-0431-y. Epub 2015 Jul 7. PMID 26149600
- [Background] Bono CM, Ghiselli G, Gilbert TJ, Kreiner DS, Reitman C, Summers JT, Baisden JL, Easa J, Fernand R, Lamer T, Matz PG, Mazanec DJ, Resnick DK, Shaffer WO, Sharma AK, Timmons RB, Toton JF; North American Spine Society. An evidence-based clinical guideline for the diagnosis and treatment of cervical radiculopathy from degenerative disorders. Spine J. 2011 Jan;11(1):64-72. doi: 10.1016/j.spinee.2010.10.023. PMID 21168100